CLINICAL TRIAL: NCT02474745
Title: Effect of the Type of Maternal Pushing During the Second Stage of Labor on Obstetric and Neonatal Outcome: a Multicenter Randomized Trial
Brief Title: Study of the Type of Pushing at Delivery
Acronym: EOLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0238; 2014-A01920-47 (Registry Identifier: 2014-A01920-47)
Record Dates: First submitted 2015-06-05; First posted 2015-06-18 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Delivery; 2nd Stage of Labor
Keywords: second stage of labor; pushing techniques

ARMS (2):
- INTERVENTION GROUP (Experimental): Directed open-glottis pushing (with prolonged exhalation) must be explained to the women and professionals as follows:
  "After inhaling deeply, the patient will exhale while pulling in her stomach in such a way they she can use the contraction of her abdominal muscles to help the fetus descend through the birth control. She should push as long as possible
  Interventions: Procedure: - Directed open-glottis pushing
- CONTROL GROUP (Other): Directed closed-glottis pushing (pushing while holding one's breath) should be explained to the women and professionals as follows:
  "After inhaling deeply, the patient should push very hard downwards to the perineum, while holding the inhaled breath in her lungs. She should push as hard and as long as possible."
  Interventions: Procedure: Directed closed-glottis pushing

INTERVENTIONS:
Procedure: - Directed open-glottis pushing — Description of the intervention in the intervention group: Directed open-glottis pushing (with prolonged exhalation) must be explained to the women and professionals as follows:
  "After inhaling deeply, the patient will exhale while pulling in her stomach in such a way they she can use the contraction of her abdominal muscles to help the fetus descend through the birth control. She should push as long as possible"
  Description of the intervention in the control group: Directed closed-glottis pushing (pushing while holding one's breath) should be explained to the women and professionals as follows:
  "After inhaling deeply, the patient should push very hard downwards to the perineum, while holding the inhaled breath in her lungs. She should push as hard and as long as possible."
  Arms: INTERVENTION GROUP
Procedure: Directed closed-glottis pushing — Description of the intervention in the intervention group: Directed open-glottis pushing (with prolonged exhalation) must be explained to the women and professionals as follows:
  "After inhaling deeply, the patient will exhale while pulling in her stomach in such a way they she can use the contraction of her abdominal muscles to help the fetus descend through the birth control. She should push as long as possible"
  Description of the intervention in the control group: Directed closed-glottis pushing (pushing while holding one's breath) should be explained to the women and professionals as follows:
  "After inhaling deeply, the patient should push very hard downwards to the perineum, while holding the inhaled breath in her lungs. She should push as hard and as long as possible."
  Arms: CONTROL GROUP

SUMMARY:
The objective of this randomized clinical trial is to assess and compare the effectiveness of directed closed-glottis (Valsalva) pushing (pushing while holding one's breath) vs. directed open-glottis pushing (pushing during a prolonged exhalation) during the second stage of labor. The study hypothesis is that open-glottis pushing results in better maternal and neonatal outcomes, in particular for maternal pelvic floor and continence function.

DETAILED DESCRIPTION:
This is a multicenter randomized, clinical trial: directed closed-glottis pushing (pushing while holding one's breath) vs. directed open-glottis pushing (pushing during a prolonged exhalation) during the active phase of labor during which the fetus descends through the birth canal (second stage).

Study plan and procedures:

During prenatal care visits, women will be informed about the study by posters hung in maternity units and midwives' offices.

All participating staff - that is, all professionals teaching childbirth preparation and parenthood classes who agree to participate in the study and midwives, who will include and randomize the women and will then manage the delivery -- will be trained in advance in both pushing techniques so that they can teach and support the women. A video intended specifically for professionals will be produced for the study and will make it possible to standardize the instruction that the professionals provide the women about each type of pushing.

Midwives (both hospital-based and in private practice) who lead childbirth preparation and parenthood classes will inform women of the study's existence. During one class session, pregnant women will receive structured instruction, including a video specifically created for the women in the study, describing both types of directed pushing. They will also have access to this training video, which will be available online at the website of the Auvergne perinatal health network (https://www.auvergne-perinat.org/). They will also receive a written brochure about the study.

Moreover, those who have completed this instruction will receive a card attesting to this instruction, which they will be asked to keep with their blood group cards (to minimize the possibility of losing it). This information will also be included in their paper obstetrics records and in their electronic records, in the section "action to be taken."

The midwives performing this instruction will provide the local study coordinator with a list of the women who were trained in these types of pushing and plan to participate in the study and to give birth in one of the participating maternity units. These lists will be available at each unit, in the study file where the information form and blank consent forms are stored.

At admission, the midwife-investigator managing the delivery will verify each woman's eligibility, inform her again about the study, and have her sign the written consent.

The co-interventions (analgesia, oxytocin, position maternal, etc.) associated with labor and its monitoring will be identical to the usual management in the participating maternity units. The midwife managing the delivery will determine the moment that active labor and thus bearing down and pushing efforts begin. In accordance with standard practice in French maternity units, clinical examination will be privileged; a preliminary ultrasound will not be performed unless otherwise planned. Nonetheless, the fetal heart rate and the frequency of uterine contractions will be monitored continuously, with an external tocodynamometer, throughout labor and expulsive efforts (no intermittent auscultation authorized after determination of eligibility/inclusion).

Investigators who determine after 20 minutes that the type of pushing used appears ineffective can ask mothers to switch to the other type, if they think it useful. In the latter case, the women will remain in their initial group (intention-to-treat analysis) but the intervention will be considered as a failure for them.

If fetal heart rate abnormalities or other obstetric emergencies occur, the midwife and/or the supervising obstetrician will be the sole decision-makers, jointly with the mother, to the extent possible for the ensuing medical management (change in pushing technique, instrumental delivery, or cesarean).

In this case, the reason for the decision will be described in the research file.

After the delivery, the midwife supervising the delivery will complete a simple descriptive form reporting adherence to the assigned pushing technique and the course of the delivery. Values for the other covariables relevant to the study will be completed by a clinical research assistant.

The women will receive a questionnaire by e-mail about her satisfaction with the management of her delivery 4 weeks afterwards. They will also be seen for a postnatal visit, mandatory in France, 6 to 8 weeks after delivery. This visit will include an examination of the pelvic floor. Women will also complete a questionnaire.

Randomization After the midwife-investigator has verified the inclusion and inclusion criteria and collected the signed informed consent, she will contact the study website and run the randomization program to allocate the woman to one of the pushing groups, according to the list described below. Once the randomization is performed, the patient will be informed of the group to which she is assigned: " open-glottis pushing" or " closed-glottis pushing". The type of pushing assigned will be used once the patient is instructed to push.

The randomization list is being created by a computer program designed by a group independent of the clinical research center and of the investigator-coordinator. It is stratified by maternity ward, according to both parity (nulliparas vs multiparas) and epidural analgesia use at randomization, and by blocks of 4 to 6. The randomization and the data collection will be performed at a website available 24 hours a day, by the investigator. Because each department has internet access either in the delivery room or the medical offices or both, this mode of randomization is possible and secure.

Data collection :

The electronic case report file (CRF) will include several parts:

* One with administrative information (center number, patient and investigator names, etc.)
* One part containing the clinical and other relevant data available in the women's medical files
* A short section to collect medical data not usually available in patient records (type of pushing, change of type of pushing, number of pushes per contraction, etc.)
* A patient satisfaction questionnaire for the women to complete
* Data related to pelvic floor status (questionnaire and clinical examination) at the postnatal check-ups after each delivery.

Before randomization, the inclusion and exclusion criteria will be verified with the aid of computer software. This computer software will also be used for all the others variables useful for this research. The randomization will take place online, at the study website. The study will not be double- or single-blinded.

The midwife-investigator managing the delivery will complete a simple descriptive form including data not usually found in patient medical records (type of pushing, number of pushes per contraction, compliance to allocated intervention).

The patients included in the study will provide their addresses, telephone numbers, and email addresses in the consent form. Should the satisfaction questionnaire not be returned after a reminder by email, she will receive a reminder by telephone.

Appointments for the postnatal check-up (study of pelvic floor function) will be made in the department before the woman's discharge. She will receive a "reminder" SMS before the appointment as well as a telephone reminder if she fails to keep the appointment. This is a mandatory postpartum consultation for all French parturients (at 6 to 8 weeks postpartum).

The study will use several different data sources:

After the delivery, the midwife-investigator will enter data for a special section of the CFR, providing information generally not included in patient medical records (adherence, station at onset of the active second stage, type of pushing, etc.) at the study website.

The patient's medical records, for most of her data. Data other than that mentioned above will be routinely collected from the medical records and reentered on the computerized study file, available at the website.

The satisfaction questionnaire will be completed online directly by the woman. The report of the postnatal check-up will similarly be entered online directly by the professional who performed it, and the questionnaire about the woman's functional perception of her pelvic floor function will be transcribed online at the same time.

Quality assurance plan :

Data collection notebook for the study:

All of the information required by the protocol must be entered into the electronic CRF. The relevant information will be recorded as it is obtained and transcribed clearly and legibly into the electronic notebook.

This electronic data collection notebook has built-in quality control features to ensure the quality of the data entry. This electronic record will be available by secure access on the website, so that the investigator-coordinator can remotely oversee the records of the maternity units participating in the study.

Moreover:

* The investigator undertakes to conduct this study in compliance with Good Clinical Practices and French public health law [Act n°2004-806 dated 9 August 2004 concerning biomedical research, its implementing decree n° 2006-477 dated 26/04/2006, which modifies the portion of the Public Health Code (specifically, Part 1, Book 1, Title II, Section 1) concerning biomedical research, as well as the decrees in force]. The investigator also undertakes to conduct this research in accordance with Declaration of Helsinki of the World Medical Association (Tokyo 2004, as revised).
* The investigator coordinator appointed by the sponsor will ensure the appropriate performance of the study, of the collection of data generated in writing, their documentation, recording, and reporting, in accordance with the standard operating procedures of the Clermont-Ferrand University Hospital Center and in compliance with Good Clinical Practices and with the applicable legislative and regulatory provisions.

The investigators guarantee the authenticity of the data collected in this study and accept the legal provisions authorizing the study sponsor to set up quality control procedures. The investigator-coordinator and all other investigators therefore agree to make themselves available for quality control inspections that will be conducted at regular intervals in the maternity units, by the investigator-coordinator. During these visits, the following items will be checked:

* Informed consent
* Compliance with the research protocol and the procedures defined therein
* Assurance of the quality of the data collected in the electronic CRF: accuracy, missing data, consistency of the data with the source documents (such as paper and electronic medical files and questionnaires completed by the midwives).

Reporting for adverse events :

According to current scientific data, conformity with the exclusion criteria for the study will ensure the lack of any threat to the life of mother or child. Pushing is an essential practice for vaginal deliveries and is a part of routine care. The data in the literature show no serious maternal or neonatal complications associated with a particular type of pushing.

Nonetheless, any serious event for mother or child, specifically transfer to an intensive care unit or death, will be reported immediately on a special form brought immediately to the attention of the principal investigator and the Sponsor.

Sample size assessment :

Based on a French national database (Audipog: http://www.audipog.net)./interro-choices.php) and on the compliance to the type of pushing found in the literature, the investigators estimate:

* For α = 0.05 and a power of 90%,
* And estimating from the Audipog database that women who deliver spontaneously, without perineal lesion (that is, without episiotomy or spontaneous 2nd, 3rd, or 4th degree lacerations) account for 49.6% of all parturients, the investigators estimate that use of a bilateral test to show an absolute difference between groups of 20% (or 49.6% vs. 69.6%, a relative difference on the order of 40%) would require 125 women per group.

Statistical analysis plan The analysis of the primary outcome will include all women who were randomized and assigned to the interventional (directed open glottis pushing) or the control group (directed closed-glottis pushing) according to an intention-to-treat analysis.

Women who did not use the type of pushing initially allocated to them by randomization will remain in their initial group for the analysis; this type of pushing will be considered a failure for them.

The potential deviations from the pushing protocol assigned and their reasons (patient's refusal or inability to follow that type, its inefficacy, clinical necessity, etc.) will be described. Ineligible inclusions should not occur, given the randomization after completion of an electronic CRF and the late point of inclusion.

The characteristics of the women included in the study will be first described. Their initial comparability will be described, especially for social and demographic data, prognostic and risk factors for our outcome measures, to take them into account with potential confounding factors in the statistical analysis.

A secondary per protocol analysis is planned.

Statistical techniques The baseline characteristics of the women and children (age, weight, parity, etc.) in the two groups will be compared with a Chi 2 test (or Fisher's exact test when appropriate) for the qualitative variables and by Student's t test for the quantitative variables.

The principal results will be reported as crude relative risks (RR) with their 95% confidence intervals. Simple descriptive statistics will be used to report some relative infrequent data (such as transfer to the NICU). A multivariate analysis (manual backward stepwise logistic regression) will be performed to take the prognostic and confounding factors into account to obtain the adjusted RRs. A center effect will be sought and handled, if necessary, with a Cochran-Mantel Haenszel test, to compare the efficacy of the type of pushing in each group An analysis according to parity is planned. Each secondary endpoint will undergo an analysis identical to that of the principal endpoint. The results will be reported as crude risks relative (RR) with their 95% confidence intervals.

An interim analysis will be planned to assess the need to adjust the study calendar. This interim analysis will be performed after half of the planned subjects have been included. Adherence to the type of pushing in France is currently unknown. To preserve an overall threshold of 5% for the final analysis, the interim analysis will use a threshold of 0.1%.

Plan for missing data The missing data will be treated as missing.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be women:
* who are nulliparas or multiparas (≥ 1 previous child),
* who attended the complete training session on the types of pushing assessed in this trial; during prenatal childbirth preparation and parenthood classes (regardless of the type of prenatal preparation)
* for whom a vaginal delivery was planned at the end of pregnancy,
* admitted to the maternity ward between 37 and 42 weeks of gestation (≥ 37 weeks and ≤ 42 weeks) in spontaneous or induced labor,
* with cervical dilatation ≥ 7 cm,
* with a singleton pregnancy in cephalic presentation,
* who provided informed consent in writing
* and speaks and writes French.

Exclusion Criteria:

* Women who are :
* minors,
* adults but incapable of providing consent for the study,
* with a disorder contraindicating prolonged pushing,
* with a uterine scar (previous cesarean or other surgery),
* with a contraindication to vaginal delivery,
* with a maternal disease that could justify in the short-term termination of the pregnancy (HELLP syndrome, preeclampsia [hypertension with albuminuria > 0.3 g by 24 hours], eclampsia, abruptio placentae, etc.),
* with a major genital hemorrhage,
* with a major fetal malformation and/or hydramnios or oligohydramnios, and/or FGR (<5°percentile), diagnosed in utero,
* with a fetal heart rate anomaly before randomization,
* with an in utero fetal death,
* with a multiple pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
composite criterion: spontaneous delivery without perineal lesion | at day 1
  (episiotomy, spontaneous 2nd, 3rd or 4th degree lacerations).

SECONDARY OUTCOMES:
occurrence of perineal lesions such as episiotomy or a severe perineal laceration | at day 1
immediate postpartum hemorrhage | at day 1
effect on pelvic floor and urinary function (POP-Q and ICIQ-SF) | at 2 months after delivery or at the postpartum visit
women's satisfaction by a Swiss validated questionnaire | at 4 weeks postpartum
  women's satisfaction at 4 weeks postpartum by a Swiss validated questionnaire (QEVA questionnaire: not yet published).

CONTACTS AND LOCATIONS:
Overall Officials: Chloé BARASINSKI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Barasinski C, Debost-Legrand A, Savary D, Bouchet P, Curinier S, Vendittelli F. Does the type of pushing at delivery influence pelvic floor function at 2 months postpartum? A pragmatic randomized trial-The EOLE study. Acta Obstet Gynecol Scand. 2023 Jan;102(1):67-75. doi: 10.1111/aogs.14461. Epub 2022 Nov 9. PMID 36352788
- [Derived] Barasinski C, Vendittelli F. Effect of the type of maternal pushing during the second stage of labour on obstetric and neonatal outcome: a multicentre randomised trial-the EOLE study protocol. BMJ Open. 2016 Dec 20;6(12):e012290. doi: 10.1136/bmjopen-2016-012290. PMID 27998899